CLINICAL TRIAL: NCT01333865
Title: A Study of Memantine Hydrochloride (Namenda®) for Cognitive and Behavioral Impairment in Adults With Autism Spectrum Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Clinical Investigator, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-000016
Record Dates: First submitted 2010-11-19; First posted 2011-04-12 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorders
Keywords: Memantine; Namenda; Autism Spectrum Disorders; Pervasive Developmental Disorders; Adults
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Namenda) Treatment (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Memantine (Namenda®) was approved by the U.S. Food and Drug Administration in 2003 and by the European Agency for the Evaluation of Medical Products in 2002 for the treatment of moderate to severe Alzheimer's disease. Evidence from available treatment trials of memantine in ASD and non-ASD populations of youth and adults strongly suggest that memantine could be an effective agent for the treatment of adults with ASD.
  During the 12 weeks of study duration, subjects will be evaluated at weekly intervals for the first 4 weeks and thereafter every 3 weeks. Memantine will be administered in divided dose twice a day in the morning and evening. Titration of study medication will be guided by a forced titration schedule with an option for slower titration or holding at lower dose per clinician judgment. Safety, effectiveness, response and side effects will be evaluated.
  Other Names: Namenda

SUMMARY:
The main objective of this study is to evaluate the safety and effectiveness of memantine (Namenda®) for cognitive and behavioral impairment in adults ages 18-50 years with autism spectrum disorders (ASD). This is an exploratory, 12-week, pilot study, seeking to determine whether Namenda is efficacious and well tolerated in the treatment of adults with ASD. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusions

* Male and female outpatients 18-50 years of age.
* Participants must have DSM-IV-TR diagnosis of PDD and displaying PDD symptoms with at least moderate impairment (SRS score ≥ 85 and CGI-PDD ≥ 4).
* Fulfills diagnosis of autism spectrum disorders by meeting DSM-IV-TR PDD diagnostic criteria of autistic disorder (with the exception of a total lack of spoken language), Asperger's disorder, or PDD-NOS as established by clinical interview and confirmed by DICA-R PDD module.
* Subjects and/or their legal representative must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Subjects and/or their legal representative must be considered reliable reporters.
* Each subject and/or their authorized legal representative must understand the nature of the study. The subject and/or their legal representative must sign an informed consent document.
* Subject must be able to participate in mandatory blood draws.
* Subject must be able to swallow pills.
* Subjects with mood, anxiety, or disruptive behavior disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.

Exclusions

* IQ < 85.
* Total lack of spoken language.
* DSM-IV-TR PDD diagnoses of Rett's disorder, or childhood disintegrative disorder.
* Clinically unstable psychiatric conditions or judged to be at serious suicidal risk.
* Active symptoms of anorexia or bulimia nervosa
* Current diagnosis of a psychotic disorder or unstable bipolar disorder.
* History of recent or current (past 30 days) clinically significant depressive or anxiety disorder that warrants treatment.
* Current diagnosis of schizophrenia.
* History of substance use (except nicotine or caffeine) within past 3 months
* Serious, stable or unstable systemic illness including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* Subjects with severe hepatic impairment (LFTs > 3 times ULN) and those with severely impaired renal function (eGFR < 30).
* Subjects with genitourinary conditions that raise urine pH (e.g., renal tubular acidosis, severe infection of the urinary tract).
* Uncorrected hypothyroidism or hyperthyroidism.
* Subjects with untreated and/or unstable diabetes.
* Non-febrile seizures without a clear and resolved etiology.
* Pregnant or nursing females.
* Known hypersensitivity to memantine.
* Severe allergies or multiple adverse drug reactions.
* A non-responder or history of intolerance to memantine, after treatment at adequate doses as determined by the clinician.
* Investigator and his/her immediate family defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by local print and Internet advertising. Participants were also recruited from the referral pool of patients in the Pediatric Psychopharmacology Program at the MGH and from the Alan and Lorraine Bressler Clinic and Research Program for ASDs.
Groups:
- Memantine (Namenda) Treatment: Memantine: Memantine (Namenda®) was approved by the U.S. Food and Drug Administration in 2003 and by the European Agency for the Evaluation of Medical Products in 2002 for the treatment of moderate to severe Alzheimer's disease. Evidence from available treatment trials of memantine in ASD and non-ASD populations of youth and adults strongly suggest that memantine could be an effective agent for the treatment of adults with ASD.
  During the 12 weeks of study duration, subjects were evaluated at weekly intervals for the first 4 weeks and thereafter every 3 weeks. Memantine was administered in divided dose twice a day in the morning and evening. Titration of study medication was guided by a forced titration schedule with an option for slower titration or holding at lower dose per clinician judgment. Safety, effectiveness, response and side effects were evaluated.
Period: Overall Study
Arm/Group | Memantine (Namenda) Treatment
Started | 19 (25 participants signed consent, but only 19 completed screening and were analyzed at baseline.)
Completed | 17 (2 participants were withdrawn. One was still analyzed, but one was withdrawn too early for analysis)
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Memantine (Namenda) Treatment: Memantine (Namenda®) was approved by the U.S. Food and Drug Administration in 2003 and by the European Agency for the Evaluation of Medical Products in 2002 for the treatment of moderate to severe Alzheimer's disease. Evidence from available treatment trials of memantine in ASD and non-ASD populations of youth and adults strongly suggest that memantine could be an effective agent for the treatment of adults with ASD.
  During the 12 weeks of study duration, subjects were evaluated at weekly intervals for the first 4 weeks and thereafter every 3 weeks. Memantine was administered in divided dose twice a day in the morning and evening. Titration of study medication was guided by a forced titration schedule with an option for slower titration or holding at lower dose per clinician judgment. Safety, effectiveness, response and side effects were evaluated.
Arm/Group | Memantine (Namenda) Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in ASD Symptom Severity as Defined by the Social Responsiveness Scale (SRS)
Description: Number of participants with reduction in ASD symptom severity defined as a reduction in Social Responsiveness Scale (SRS) score from baseline of greater than or equal to 30%.
  The SRS is a 65-item rating scale completed by an informant to measure the severity of autism spectrum symptoms as they occur in natural settings.
Time Frame: Week 12
Population: 19 participants were exposed to the medication, but 1 withdrew due to feeling mildly sedated which affected his driving. This occurred too early in the study for him to be analyzed.
Measure: Number; unit: participants
Arm/Group | Memantine (Namenda) Treatment
Number analyzed (Participants) | 18
participants | 6

2. Secondary Outcome: Number of Participants With Reduction in ASD Symptom Severity as Defined by the NIMH Clinical Global Impression for Pervasive Developmental Disorders (CGI-PDD) Improvement Score
Description: Number of participants with reduction in ASD symptom severity defined as an NIMH Clinical Global Impression (CGI) Pervasive Developmental Disorder (PDD) Improvement score less than or equal to 2. The CGI-Improvement is a clinician-rated measure of improvement. Scores range from 1 (very much improved) to 7 (very much worse) for PDD.
Time Frame: Pre-treatment - 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Memantine (Namenda) Treatment
Number analyzed (Participants) | 18
participants | 15

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Memantine (Namenda) Treatment: Memantine (Namenda®) was approved by the U.S. Food and Drug Administration in 2003 and by the European Agency for the Evaluation of Medical Products in 2002 for the treatment of moderate to severe Alzheimer's disease. Evidence from available treatment trials of memantine in ASD and non-ASD populations of youth and adults strongly suggest that memantine could be an effective agent for the treatment of adults with ASD.
  During the 12 weeks of study duration, subjects were be evaluated at weekly intervals for the first 4 weeks and thereafter every 3 weeks. Memantine was administered in divided dose twice a day in the morning and evening. Titration of study medication was guided by a forced titration schedule with an option for slower titration or holding at lower dose per clinician judgment. Safety, effectiveness, response and side effects were evaluated.
Arm/Group | Memantine (Namenda) Treatment
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 14/19
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (Namenda) Treatment (N=19)
Sore Throat (General disorders) | 1 (2)
Decreased appetite (General disorders) | 2 (2)
Headache (General disorders) | 4 (8)
Dizziness (General disorders) | 3 (3)
Lower jaw pain (General disorders) | 1 (1)
PMS symptoms (General disorders) | 1 (1)
Severe meltdown (General disorders) | 1 (1)
Depressed mood (General disorders) | 2 (2)
Insomnia (General disorders) | 4 (5)
Nausea (General disorders) | 1 (1)
Tiredness/sedation (General disorders) | 7 (7)
Back pain (General disorders) | 2 (2)
Dissociated/emotionless (General disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
Common cold/sinus (General disorders) | 2 (3)
Left food pain/tingling (General disorders) | 2 (2)
Kidney stone pain (General disorders) | 1 (1)
Lighteheaded (General disorders) | 2 (2)
Decreased sex drive (General disorders) | 1 (3)
Dysmenorrhea (General disorders) | 1 (1)
Burning in urine (General disorders) | 1 (1)
Mispronouncing words (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes